CLINICAL TRIAL: NCT00698360
Title: Circadian Rhythm of Erythropoietin and Melatonin in Patients With Various Degrees of Renal Insufficiency
Brief Title: Circadian Rhythm of Erythropoietin And Melatonin in Renal Disease
Acronym: CREAM 1
Status: Completed | Type: Observational
Sponsor: Meander Medical Center (Other)
Collaborators: Stichting Bijstand, Meander Medical Center (Unknown); Hoffmann-La Roche (Industry)
Responsible Party: Meander Medical Center
Other Study IDs: CREAM 1; R-07.03M
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; melatonin; erythropoietin; circadian rhythm
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- A: MDRD 10-30
- B: MDRD 30-60
- C: MDRD 60-80
- D: MDRD > 80

SUMMARY:
Rationale: Investigation of the circadian rhythm of erythropoietin and melatonin in patients with various degrees of renal insufficiency

Objectives:

Primary objective: Is there a circadian rhythm of epo and melatonin in patients with various degrees of renal insufficiency?

Primary Objective: Is there a circadian rhythm of epo and melatonin in patients with various degrees of renal insufficiency compared to patients with a normal renal function?

Secondary Objective: Is there a circadian rhythm of cortisol and IGF in patients with various degrees of renal insufficiency?

Secondary Objective: Is there a circadian rhythm of cortisol and IGF in patients with various degrees of renal insufficiency compared to patients with a normal renal function?

Study design: Comparative study in 4 groups with various degrees of renal insufficiency, duration for each patient 24 hrs. Total duration of study 12 months, patients admitted to the hospital (on nursing ward)

Study population: Patients with various degrees of renal insufficiency

Main study parameters/endpoints: Analysis of the existence of a circadian rhythm in patients with a normal renal function and in patients with variable degrees of renal insufficiency

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Better knowledge of the circadian rhythm in renal insufficiency. This could lead to a more efficient administration of erythropoietin and melatonin in the future.

Extent of burden is 1 venapunction for placement of infusion needle, the withdrawal of 11 times 5 ml blood in 24 hrs, continuous measurement of body temperature via capsule, 24-hour continuous ambulant blood pressure monitoring.

ELIGIBILITY:
Inclusion criteria:

* Patient with various degrees of renal insufficiency, stable creatinin clearance: minimum 10 ml/min (measured with MDRD), admitted to our hospital
* Informed Consent
* Man/Women between 18 and 85 years
* Understanding and knowledge of the dutch language

Exclusion criteria:

* Instable angina pectoris, heart failure NYHA class IV
* Therapy with erythropoetin, melatonin and hypnotics
* Acute renal failure or rapidly progressive glomerulonephritis
* Bleeding or hemolysis as a cause of anemia
* Deficiency of iron, folate and/or vitamin B12
* Presence of chronic inflammatory disease or clinically significant infection
* Hemoglobinopathies
* Alcohol and/or drug abuse
* Enrolment in another study
* Any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with various degrees of renal insufficiency, admitted to Meander Medical Center
  * A: Patients with renal insufficiency (clearance 10-30 ml/min)
  * B: Patients with renal insufficiency (clearance 30-60 ml/min)
  * C: Patients with renal insufficiency (clearance 60-80 ml/min)
  * D: Patients with normal renal function (clearance > 80 ml/min)
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2007-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
existence of circadian rhythm of Erythropoietin and Melatonin | 24 hours

SECONDARY OUTCOMES:
existence of a circadian rhythm of cortisol and IGF-1 | 24 hours
Relationship between temperature and melatonin. Relationship between blood pressure and erythropoietin | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Carlo AJM Gaillard, MD PhD, Study Chair — Meander Medical Center
Locations (1):
- Meander Medical Center, Amersfoort, Netherlands